CLINICAL TRIAL: NCT07062861
Title: Comparison of Proximal and Distal Cannulation of the Radial Artery by Ultrasonography in Pediatric Patients Undergoing Elective Surgery
Brief Title: Proximal and Distal Radial Artery Cannulation in Children
Status: Recruiting | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assoc. Prof., Marmara University
Other Study IDs: 09.2025.25-0131
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-07

CONDITIONS: Arterial Catheterization; Radial Atrery Cannulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group P: Radial arterial cannulation from the proximal part of the artery.
- Group D: Radial arterial cannulation from the distal part of the artery.

SUMMARY:
Intraarterial cannulation is important for continuous blood pressure monitoring and blood gas analysis throughout the surgical procedure and in intensive care patients. Ultrasonography (USG) has gained popularity in vascular cannulations and facilitates intraarterial interventions. Radial artery is one of the most preferred arteries. Our aim in this study is to compare proximal and distal radial artery cannulations by USG in pediatric patients in terms of procedural success, procedure time and complications.

DETAILED DESCRIPTION:
After the patients are admitted to the operating room, routine monitoring (electrocardiography, noninvasive blood pressure and peripheral oxygen saturation) will be performed. After appropriate vascular access is provided to the patients, the induction phase of general anesthesia will begin. Anesthesia induction will be left to the choice of the primary anesthesiologist and no protocol will be followed. In case of >25% drop in blood pressure, 0.1 mcg/kg noradrenaline will be administered intravenously. After the appropriate position is given to the arm of the patient to be treated, radial artery cannulation will be performed with USG obeying asepsis rules. Patients will be divided into 2 groups. The first group will be the patients who will be cannulated at the level of the distal radius (styloid process). For the second group, proximal radial artery cannulation will be performed proximally from the styloid process by measuring 1 cm in patients under 20 kg, 2 cm between 20-30 kg, 3 cm between 30-40 kg, 4 cm between 40-50 kg, and 5 cm in patients over 50 kg. Demographic and clinical characteristics of the patients will be recorded. Catheterization success rates, procedure duration, number of interventions, vessel diameter, hematoma at the site of intervention on the 1st postoperative day, circulatory disturbance will be examined.

ELIGIBILITY:
Inclusion Criteria:

* PEDIATRIC patients undergoing elective surgery
* ASA I-III physical status

Exclusion Criteria:

* Refusal to participate in the study
* Those with peripheral vascular disease
* Vasopressor drug users
* Infection or anatomical defects at the site of the procedure
* Patients with coagulation disorders

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients aged 4-14 years undergoing elective surgery under general anesthesia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Success rate | From the preinduction period in the operating theater to the postoperative day one.
  Radial artery catheterization success rates will be compared between the groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Will be decided at the end of the study.